CLINICAL TRIAL: NCT02727933
Title: Postmarketing Surveillance of the Safety and Effectiveness of Daclatasvir and Asunaprevir for the Treatment of Chronic HCV Genotype 1B Infection in the Routine Clinical Practice in Korea
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI444-335
Record Dates: First submitted 2016-03-18; First posted 2016-04-05 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to describe the safety of the combination of Daklinza (daclatasvir) and Sunvepra (asunaprevir) when used for the treatment of chronic hepatitis C (CHC) genotype 1b patients in real-life conditions when used according to its registered indications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CHC genotype 1b and compensated liver disease, including cirrhotic patients
* Eligible for treatment with Daklinza and Sunvepra as indicated in the locally approved prescribing information.

Exclusion Criteria:

* Off-label use of Daklinza and Sunvepra
* Patients with a contraindication for the use of Daklinza and Sunvepra as described in the locally approved prescribing information

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 1941 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2020-07-05 (Actual); Study Completion 2020-07-05 (Actual)

PRIMARY OUTCOMES:
Frequency of expected and unexpected adverse reactions (AEs) and serious adverse events (SAEs)/reactions. These include laboratory abnormalities | 6 months to 5 years

SECONDARY OUTCOMES:
Incidence proportion of AEs leading to discontinuation of study therapy | 6 months to 5 years
Incidence rate of AEs leading to discontinuation of study therapy | 6 months to 5 years
Timing of laboratory abnormalities by toxicity grade | 6 months to 5 years
Percentage of patients with HCV (Hepatitis C Virus) RNA (Ribonucleic acid)< lower limit of quantification (LLQ) target not detected and detected | 4 Weeks to 24 Weeks
The sustained virologic response (SVR12) of the combination of Daklinza and Sunvepra (HCV RNA < lower limit of quantification [LLQ] target not detected and detected (HCV RNA < 25 IU/mL) | 24 Weeks to 36 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Seoul, South Korea

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm